CLINICAL TRIAL: NCT04931797
Title: Using the Emergency Department Visit to Promote Advance Care Planning
Brief Title: Video Images About Decisions for Ethical Outcomes in the Emergency Department (VIDEO-ED)
Acronym: VIDEO-ED
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of California, Davis (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Angelo E. Volandes, MD, Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2021p001552; R01AG065254 (NIH)
Record Dates: First submitted 2021-06-01; First posted 2021-06-18 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Outcomes Assessor
Masking Description: Primary outcome will be obtained through natural language processing (NLP) from the EHR, in which the RA conducting the NLP will not know which arm of the study the patient was in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video (Experimental): Video decision aid and advance care planning discussion
  Interventions: Behavioral: video decision aid
- Control arm (Active Comparator): Usual advance care planning services provided at the study site.
  Interventions: Behavioral: control arm ACP information sheet

INTERVENTIONS:
Behavioral: video decision aid — advance care planning video decision aid
  Arms: Video
Behavioral: control arm ACP information sheet — control arm ACP information sheet
  Arms: Control arm

SUMMARY:
A randomized controlled trial of a video decision aid in the Emergency Department Setting to improve advance care planning documentation.

DETAILED DESCRIPTION:
A randomized controlled trial of a video decision aid in the Emergency Department setting shown to patients followed by a brief advance care planning discussion and then relay that discussion to the patient's primary care provider and/or admitting clinical team and look at rates of advance care planning documentation in the electronic health record over time. Primary outcome is advance care planning documentation in the EHR at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* anyone aged 65 and over or anyone aged over 50-64 with an indicator of serious illness

Exclusion Criteria:

* non english or spanish speakers those with a POLST legally blind medically non stable requiring ICU level care

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
EHR documentation of advance care planning | 3 months
  EHR documentation of advance care planning

SECONDARY OUTCOMES:
patient reported conversations with health care providers and family | at 3 and 6 months
  patient reported conversations with health care providers and family
concordance between stated and documented preferences | at 3 and 6 months
  concordance between stated and documented preferences
ACP documentation in the EHR | at 6 months
  ACP documentation in the EHR
hospitalization | at 3 and 6 months
  hospitalization
differential intervention effects of the ACP video intervention on patient ACP documentation based on race and ethnicity | at baseline, 3 and 6 months
  We will look at ACP documentation in the intervention and control arms to see if there are differential intervention effects based on race and ethnicity. We will look at the ACP documentation rate in Whites in both arms, and compare them to African Americans and Latinx populations. We will be able to see if the intervention had a greater or lesser effect on ACP rates in sub groups of our population by race and ethnicity.
quality of clinician ACP communication using an ACP quality communication survey | quality of communication at the time of the survey interview (baseline), and then at 3 and 6 months
  quality of ACP communication using an ACP quality communication survey
place of death | at 3 and 6 months
  place of death
enrollment in hospice | at 3 and 6 months
  enrollment in hospice
ED visits | at 3 and 6 months
  ED visits
mortality | at 3 and 6 months
  mortality
ICU days | at 3 and 6 months
  ICU days
patient CPR and breathing machine preferences | at time of survey (baseline) and then after 3 and 6 months
  we will ask the patient whether or not they want CPR attempted and whether they would wish to be placed on a breathing machine
patient preferences for goals of care | at time of survey (baseline) and then after 3 and 6 months
  We will ask patient if they wish to receive life prolonging care, limited care or comfort care.
decisional certainty regarding decision making for ACP preferences | at baseline survey interview
  we will ask patients how certain they are about their decisions for the goals of care
patient knowledge of ACP | at baseline survey interview
  We will ask patients knowledge questions about their understanding of advance care planning
patient confidence in health care delivery that is aligned with patient preferences | at time of survey (baseline) and then after 3 and 6 months
  We will ask patients how confident they are in that they will receive the type of medical care they wish in their health care system
patient ACP engagement with ACP topics | at baseline survey interview
  We will ask patients how ready and engaged they are with the topic of advance care planning

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UC Davis, Davis, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Newton Wellesley Hospital, Newton, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: 1 year after all primary and secondary publications published.